CLINICAL TRIAL: NCT01603199
Title: Impact of a High-protein High-fiber Diet on the Nutritional Status of Patients With Primary Biliary Cirrhosis
Brief Title: High-protein High-fiber Diet in Patients With Primary Biliary Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GAS-460-11/12-1
Record Dates: First submitted 2012-05-17; First posted 2012-05-22 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary biliary cirrhosis (Non-cirrhotic) (Experimental)
  Interventions: Dietary Supplement: High protein high fiber diet
- Primary biliary cirrhosis (Cirrhotic) (Experimental)
  Interventions: Dietary Supplement: High protein high fiber diet

INTERVENTIONS:
Dietary Supplement: High protein high fiber diet — A personalized high protein high fiber dietary plan will be provided to each participant from both groups. Each participant will receive nutritional counseling once a month during six months.

SUMMARY:
Primary biliary cirrhosis is a chronic cholestatic autoimmune liver disease with a progressive course that can lead to liver cirrhosis. There are few studies on dietary management in primary biliary cirrhosis and most of them have focused on micronutrients specifically vitamin D intake to prevent osteoporosis, and lipid control to prevent hyperlipidemia, but few recommendations have been made regarding a complete dietary approach. Fiber has been proven to increase the excretion of nitrogen products and consequently reduce its blood levels, and an adequate protein intake (1- 1.5 g per kg) has shown to decrease endogenous catabolism in cirrhotic patients.

The purpose of this study is to evaluate the impact of a high-protein, high-fiber diet in the nutritional status of patients with primary biliary cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Controls

Diagnose of primary biliary cirrhosis:

* Biochemical evidence of cholestasis: based mainly on alkaline phosphatase elevation
* Presence of antimitochondrial antibodies (AMA)
* Histologic evidence of nonsuppurative destructive cholangitis and destruction of interlobular bile ducts.

Ambulatory patients

* Cases

Diagnose of primary biliary cirrhosis:

* Biochemical evidence of cholestasis: based mainly on alkaline phosphatase elevation
* Presence of antimitochondrial antibodies (AMA)
* Histologic evidence of nonsuppurative destructive cholangitis and destruction of interlobular bile ducts.

Diagnose of liver cirrhosis by two or more of the following criteria:

* Albumin < 3.4 g/dL
* INR ≥ 1.3
* Total bilirubin ≥ 2 mg/dL
* Portal hypertension (esophageal varices, splenomegaly, ascites, etc.)
* Liver biopsy Ambulatory patients

Exclusion Criteria:

* Overlapping syndrome with predominant autoimmune hepatitis
* Hospitalized patients
* Acute or chronic renal failure
* Hepatocellular carcinoma
* Pregnancy
* Neuropsychiatric disorders (Schizophrenia, bipolar disorder, dementia and attention-deficit hyperactivity disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Participants will be followed for 6 months
  Measured with the following parameters: body weight and height (to calculate BMI), triceps skinfold thickness and mid-arm circumference (to calculate mid-arm muscle circumference. Fat mass, fat free mass, total, intracellular and extracellular body water obtained by bioelectrical impedance analysis, and individual vectors obtained by bioelectrical impedance vector analysis.

SECONDARY OUTCOMES:
Minimal hepatic encephalopathy | Participants will be followed for 6 months
  Assessed by Psychometric Hepatic Encephalopathy Score (PHES) and Critical Flicker Frequency (CFF)
Quality of life | Participants will be followed for 6 months
  Assessed by SF-36 and PBC-40 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, M.D. M.Sc, Study Chair — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico